CLINICAL TRIAL: NCT00348959
Title: An Evaluation of the Effect of 'Open Window', an Art Intervention, on Psychological Well-being and Experience of Stem Cell Transplantation for the Treatment of Haematological Malignancies
Brief Title: An Evaluation of the Effect of 'Open Window' on Psychological Well-being and Experience of Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Irish Cancer Society (Other)
Responsible Party: Principal Investigator, Catherine McCabe, Research Fellow, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSY04MCC
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Hematological Malignancies
Keywords: Haematological Malignancies; Autologous Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Quality of Life; Life Threatening Illness; Art in Health Care; Randomised Controlled Trial; Mixed Methods Research
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 'Open Window' Project — Open Window' is an entirely art based intervention comprising a multimedia system that uses a combination of video projectors, audio speakers and bespoke software to make images appear as a 'virtual window' on the wall of the patients' room. Artists use mobile phone cameras and camcorders to record the images that are sent to the unit over the internet and via mobile phone networks. Original music composed for the project may also accompany the images as they appear.
  Artists are commissioned to create work for the 'Open Window' project and are aware of the nature of the viewer and the context in which the art will be shown. The art in 'Open Window' encourages the viewer to think about and engage in what they see from their own personal frame of reference.
  Other Names: Art Intervention

SUMMARY:
The 'Open Window' Study is a prospective longitudinal study using a 4 group randomised control trial design to evaluate the psychological effect of 'Open Window' on the consequences of long term isolation on patients undergoing stem cell transplantation treatment of haematological malignancies. This study uses a randomised control trial design, which is widely used in healthcare settings to test the effects of interventions and testing cause and effect relationships between variables. A mixed methods approach for data collection and data analysis is being used. This will facilitate measurement of patients' psychological response to 'Open Window' using questionnaires and exploration of subjective feelings in relation to personal experiences of having a stem cell transplant through semi structured interviews.

Hypothesis to be tested

'Open Window' has no effect on patients' levels of anxiety, depression, or distress when undergoing a stem cell transplant.

Results:

Of the 199 patients in the study, 96 were randomized to the intervention group and 103 to the control group. Participants in the intervention group had significantly reduced levels of anxiety on the day before transplant (P = 0.001), at day 7 (P = 0.041), and day 60 (P = 0.035). There was a significant reduction in depression before transplant (P= 0.022). Participants in the intervention group reported better experiences (P < 0.005).

DETAILED DESCRIPTION:
'Open Window' is a unique and novel intervention for patients being treated for haematological malignancies in the 'National Stem Cell Transplant Unit', St. James' Hospital, Dublin, Ireland. Treatment programmes include allogeneic and autologous stem cell transplantation for leukaemia and related disorders. This unit comprises 21 single air-conditioned rooms in which patients are treated and cared for. The unit is located on the ground floor of a large hospital and the view out of most of the windows is limited to the light railway system at best and the air conditioning unit at worst. Windows in the rooms are quite large although light and sunlight is limited in some by an adjacent building. The rooms vary in size and shape and all are en suite and contain a bed, locker, easy chair and TV/video mounted high on the wall, usually to the left, in front of the patient. All rooms are painted in magnolia with a blue door to the en suite and exit. In order to reduce the risk of infection, flowers and pictures hanging on the walls are prohibited and personal items such as photos are limited. Blinds are used on the windows and bed covers are blue, pink or green. The overall effect is minimalist and clinical due to the presence of medical equipment. Visiting is limited and children under 14 years of age are not allowed to visit.

Although a new unit, The National Transplant Unit was not purpose built and the focus of the design was in providing a protective environment for as many patients as possible within a limited space and with very specific requirements. While it is arguable that the introduction of colour to the walls and the inclusion of patterned curtains or bedspreads might enhance the environment from a design perspective, in the absence of such an initiative, this atmosphere provides an ideal opportunity to assess the effect of art on the experience of a very specific group of patients in a controlled atmosphere. Redshaw (2004) suggests that design alone does not provide spaces that are attractive, imaginative and engaging but that it is the inclusion of art that does this. Her study on the impact of the provision of art in a children's hospital is reported as providing a distraction for children and parents, providing enjoyment and comfort, facilitating self-expression and building self-esteem and confidence. This function of art in healthcare fulfills its role in providing a healing environment and is the primary reason why it was considered an appropriate intervention for the specific population of patients included in the 'Open Window' project.

People have a basic need for contact with each other. Isolation from people, or separation from familiar places, can cause feelings of despair, anger and hopelessness (Denton 1986; Jenner 1990; Gammon 1998). Views of nature or people through a window reduce the negative effects of isolation and can impact positively on psychological well-being (Kennedy & Hamilton 1997, Ulrich 1983). Due to the location, design and décor of the rooms, the patients in 'The National Stem Cell Transplant Unit' at St. James's have very little stimulation other than TV, radio and reading. It is arguable that a patient-centred hospital environmental design may be sufficient to make their experience more comfortable and aesthetically pleasing; however, it is the inclusion of art in the environment that may provide a more positive and enduring distraction for patients and have a positive influence on a patient's sense of 'self' and well-being and overall psychological adjustment to having a life threatening illness. This is important in providing holistic care for patients and may influence their immediate and long-term recovery.

'Open Window' is an entirely art based intervention comprising a multimedia system that uses a combination of video projectors, audio speakers and bespoke software to make images appear as a 'virtual window' on the wall of the patients' room. Artists use mobile phone cameras and camcorders to record the images that are sent to the unit over the internet and via mobile phone networks. Original music composed for the project may also accompany the images as they appear. The curator and artist in residence on the project can discuss with the patient and family, the possibility of obtaining familiar and/or family images if they wish. Patients can turn the system on, off and change the images by pressing the appropriate button on the remote control. They can also choose to include or exclude certain images if they wish. The volume of the music that accompanies some of the video channels can be controlled using the remote control.

Artists are commissioned to create work for the 'Open Window' project and are aware of the nature of the viewer and the context in which the art will be shown. The art in 'Open Window' encourages the viewer to think about and engage in what they see from their own personal frame of reference. The artist and theorist, Duchamp (1957, 3) described this process as the viewer "bringing the work in contact with the external world by deciphering and interpreting its inner qualification". These principles give patients who wish to use 'Open Window' the opportunity to become part of the creative process regardless of their past experience or knowledge of art. Patients may benefit because 'Open Window' becomes whatever they want it to be and helps them deal with their physical, psychological and social needs in a unique and individualized way.

The 'Open Window' Intervention has three aims. The first is to help patients deal with being in a restricted protective environment for 4-6 weeks. The second is to give patients a sense of connection with the outside world and the third is to provide a medium through which patients may reflect on having a life threatening illness, which may have immediate, and long-term effects on their psychological adjustment to recovering from and possibly surviving stem cell transplantation.

Results:

One hundred and ninty nine patients took part in the study, 96 were randomized to the intervention group and 103 to the control group. The intervention group had significantly reduced levels of anxiety on the day before transplant (P = 0.001), at day 7 (P = 0.041), and day 60 (P = 0.035). Participants in the intervention group reported better experiences (P < 0.005). Qualitative data showed that those in the intervention group reported that 'Open Window' was a great distraction from their illness and isolation and provided a connection with outside 'normal' life.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Denis Burkitt unit for an autologous or allogeneic stem cell transplant.

Patients who gives informed consent to participate in the study Patients who can read and speak English reasonably well. Patients who do not have communication difficulties, intellectual disabilities or known mental illness Patients who will be treated as an in-patient in the Denis Burkitt Unit following transplantation.

Exclusion Criteria:

Patients who are not undergoing a stem cell transplant Patients who do not consent to participate in the study Patients with communication difficulties, learning disabilities, mental illness, prisoners, young offenders.

Patients who are transferred to other units immediately following transplantation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are Anxiety, Depression and Distress. Measures will be taken on 7 occasions over a six month period. | Six Months

SECONDARY OUTCOMES:
Patient expectations in relation to the experience of having a stem cell transplant. | Day + 30

CONTACTS AND LOCATIONS:
Overall Officials: Shaun McCann, Study Director — St. James's Hospital, Ireland; Catherine McCabe, BNS, MSc, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St. James's Hospital, Dublin, Dublin, Ireland

REFERENCES:
- [Derived] McCabe C, Roche D, Hegarty F, McCann S. 'Open Window': a randomized trial of the effect of new media art using a virtual window on quality of life in patients' experiencing stem cell transplantation. Psychooncology. 2013 Feb;22(2):330-7. doi: 10.1002/pon.2093. Epub 2011 Dec 6. PMID 22147646
- See also: Describes human connectedness as one of the concepts underpinning this intervention — http://web.media.mit.edu/~stefan/hc/projects/openwindow/
- See also: Discusses how the 'Open Window' study demonstrates how art and science can be and possibly should be interlinked — http://seedartscience.blogspot.com